CLINICAL TRIAL: NCT04165005
Title: Mindfulness-based Short Intervention for Seniors - Decentering Effects on Cognitive Functions and Psychological Distress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Collaborators: Ruppin Acdemic Center (Other)
Responsible Party: Principal Investigator, Ophir Leshets, MA student, MA in the clinical-gerontological program, Ruppin Academic Center, Ben-Gurion University of the Negev
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 597
Record Dates: First submitted 2019-11-01; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Old Age; Debility; Psychological Distress; Cognitive Change
Keywords: elderly; MBSR; cognitive functions; psychological status
MeSH Terms: conditions — Frailty | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- decentering group (Experimental): MBSR focused on a "decentering" component (i.e. individuals observe their feelings and thoughts as ephemeral events, with no reactivity, alongside with acceptance).
  Interventions: Behavioral: decentering
- guided imagery group (Experimental): a group practicing in guided imagery sessions.
  Interventions: Behavioral: guided imagery
- control group (No Intervention): usual care group

INTERVENTIONS:
Behavioral: decentering — examined a mindfulness-based intervention focused on a decentering component, that is suitable for elders, aimed to influence on cognitive measures and psychological distress.
  Arms: decentering group
Behavioral: guided imagery — relaxing guided imagery including breathing exercises.
  Arms: guided imagery group

SUMMARY:
The present study examined the effect of a short Mindfulness-based intervention emphasizing a 'decentering' component on elderly seniors. Methods: 30 community seniors (Mage= 74.7) performed either 'decentering' intervention, guided imagery intervention, or control care as usual. The 8-week interventions included weekly 20-minute sessions and daily 10-minute home practice. Participants underwent a cognitive and emotional assessment before and after the interventions, which included filling out questionnaires and performing the Simon task. Trial registration: The study follows the principles of the Declaration of Helsinki, approved by the committee in Beer-Yaacov Hospital, Israel (number 579) on 24 Oct. 2017.

ELIGIBILITY:
Inclusion Criteria:

* age 65 and above
* membership in the study's specific enrollment community centers
* scoring 24 and above in the Mini-Mental State Examination (MMSE).

Exclusion Criteria:

* age under 65
* not being a member in the study's specific enrollment community centers
* scoring under 24 in the Mini-Mental State Examination (MMSE).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Simon task- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  a cognitive task, assessing control processes under speeded conditions, measured by response time and accuracy rate. shorter response time and higher accuracy rate indicate better performance.

SECONDARY OUTCOMES:
FFMQ- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  The Five-Fact Mindfulness Questionnaire, a manipulation check of mindfulness, ranging from 1 to 5, with higher score indicating higher mindfulness level
PWB questionnaire- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  The Psychological Well-Being Questionnaire, ranging from 1 to 6, with higher score indicating higher well-being level
MMSE- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  the Mini-Mental State examination: a cognitive function measure for elders, used to determine participation eligibility. the animation score ranges between 0 to 30, with higher score indicating better cognitive functioning
PHQ-9- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  The Patient Health Questionnaire - a depression levels measure, ranging from 0 to 3, with higher score indicating higher depression level
BDI-II- change from baseline to after intervention | at baseline and through intervention's completion, 10 weeks.
  The Beck Depression Inventory-II- a depression levels measure, ranging from 1 to 4, with higher score indicating higher depression level

CONTACTS AND LOCATIONS:
Locations (1):
- Ruppin Academic Center, Emek-Hefer, Emek-Hefer, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aisenberg-Shafran D, Shturm L. The effects of mindfulness meditation versus CBT for anxiety on emotional distress and attitudes toward seeking mental health treatment: a semi-randomized trial. Sci Rep. 2022 Nov 16;12(1):19711. doi: 10.1038/s41598-022-24256-9. PMID 36385638